CLINICAL TRIAL: NCT00581685
Title: Does Optimal Pain Control With Pregabalin and Celecoxib Predict Improved Function After Total Hip Arthroplasty?
Brief Title: Does Optimal Control of Pre-operative Chronic and Acute Pain Predict Improved Function After Orthopedic Surgery?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Dr. Colin McCartney, Staff Anesthesiologist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 216-2007; PSI-07-52
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Osteoarthritis
Keywords: Chronic pain; Preemptive analgesia; Pregabalin; Celecoxib; Hip Arthroplasty; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Chronic Pain | interventions — Pregabalin; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 (Placebo Comparator): Prospective, single center, randomized, double-blinded, placebo controlled study
  Interventions: Drug: Pregabalin, Celecoxib

INTERVENTIONS:
Drug: Pregabalin, Celecoxib — Pregabalin (75mg BID) and Celecoxib(100mg BID) two weeks prior to hip arthroplasty and 3 weeks postoperatively.

SUMMARY:
Despite the development of new pain medications, the prevalence of persistent postoperative pain (for more than three to six months) remains alarmingly high. Chronic pain and reduced function after surgery are of great concern since they have a significant impact on a patient's quality of life and are costly to society in terms of longer hospital stays and lost work days. An important risk factor for chronic pain and reduced function after surgery is the amount of pain patients experience immediately after surgery which is highly influenced by the amount of pain patients have preoperatively. For many patients, longstanding pain prior to surgery is common and thus can compromise the outcome of the procedure. Therefore, the aim of this study is to reduce the amount of pain patients have before they undergo surgery by administering a novel pain-relieving regimen in the weeks before surgery. Crucially, this treatment will be continued for three weeks after surgery to reduce pain that arises from the surgical trauma. The novel regimen will include a non-steroidal anti-inflammatory (celecoxib) and the alpha2 delta ligand, pregabalin. This drug combination will provide the best opportunity to target several key sites in the pain pathway. This regimen will be tested in patients with pain related to osteoarthritis and who are undergoing orthopedic (hip) surgery because chronic preoperative pain is common in these patients and is the main reason for undergoing surgery. The goal of this research proposal is to adequately manage pain before and after surgery in order to improve function weeks after surgery. If controlling pain in this way does lead to improved long term postoperative function the findings from this study may lead to the development of a standardized regimen. This is highly relevant not only for orthopedic procedures but following other common surgical procedures which would be of great benefit to patients and the entire healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* American Society of Anesthesiologists physical status I-III
* Average daily VAS ≥ 4
* Aged 18 - 75 years
* Male or female
* Scheduled for total hip arthroplasty (THA).

Exclusion Criteria:

* Allergy to study medications or local anesthetics
* History of drug or alcohol abuse
* Patients with chronic pain on slow-release preparations of opioid (>30mg morphine equivalent per day)
* Patients with rheumatoid arthritis
* Patients with psychiatric disorders
* Patients unable or unwilling to use Patient Controlled Analgesia (PCA).
* Diabetic patients or those with impaired renal function (Creatinine > 55)
* Obese patients (i.e. BMI > 40).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Physical function | 6 weeks postop

SECONDARY OUTCOMES:
Pain | Pre and postoperatively (up to 6 weeks)